CLINICAL TRIAL: NCT05933512
Title: A Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01E-2 (COVID-19 Beta/Omicron (BA.1/BQ.1.1/XBB.1) Variants S-Trimer Vaccine) in Population Previously Vaccinated With mRNA COVID-19 Vaccine
Brief Title: A Study to Evaluate the Immunogenicity and Safety of A Recombinant Protein COVID-19 Vaccine as Booster Vaccines
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01E-2-CHN-1
Record Dates: First submitted 2023-07-04; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: SARS-CoV-2; COVID-19; vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group A was designed as double-blinded and Group B was open label.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:SCTV01E-2 (Experimental): one dose of SCTV01E-2 on D0
  Interventions: Biological: SCTV01E-2
- Group A:SCTV01E (Active Comparator): one dose of SCTV01E on D0
  Interventions: Biological: SCTV01E
- Group B:SCTV01E-2 (Experimental): one dose of SCTV01E-2 on D0
  Interventions: Biological: SCTV01E-2

INTERVENTIONS:
Biological: SCTV01E-2 — intramuscular injection
  Arms: Group A:SCTV01E-2; Group B:SCTV01E-2
Biological: SCTV01E — intramuscular injection
  Arms: Group A:SCTV01E

SUMMARY:
This study is a phase Ⅱ clinical trial to evaluate the safety and immunogenicity of SCTV01E-2 in people of different ages who had been vaccinated with COVID-19 vaccines. A total of at least 600 subjects aged 3 years and older who were previously vaccinated with domestically licensed SARS-CoV-2 vaccines with recommended doses and immunization schedules are planned to be enrolled. Group A included 400 patients aged 18 years and above, and group B included 200 patients aged 3-17 years.

DETAILED DESCRIPTION:
For participants in Group A, they will be randomized to receive SCTV01E or SCTV01E-2 in a ratio of 1:1. For participants in Group B, they will all receive SCTV01E-2.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged ≥3 years old when signing ICF;
* 2. Participants who were vaccinated with licenced COVID-19 vaccines with recommended doses and immune schedule, and the interval between the last dose and ICF is ≥6 months.
* 3. The participant and/or his/her legal guardians or entrusted person can sign the written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
* 4. The participant and/or his/her legal guardians or entrusted person have the ability to read, understand, and fill in record cards;
* 5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
* 6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

* 1. Presence of fever within 72 hours before the study vaccination (for participants >14 years old, axillary temperature ≥37.3℃; for participants ≤14 years old, axillary temperature ≥37.5℃;);
* 2. A positive result of antigen test or nucleic acid test for SARS-CoV-2 during the screening period;
* 3. A positive result of SARS-CoV-2 IgM test;
* 4. Known history of SARS-CoV-2 infection within 6 months before ICF;
* 5. A history of sereve allergic reactions such as severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema, or allergic reactions to the study vaccines and its ingredient;
* 6. A medical or family history of seizure, epilepsy and psychosis;
* 7. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
* 8. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
* 9. Patients on antituberculosis therapy;
* 10. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
* 11. Participants who received other investigational drugs within 1 month before the study vaccination;
* 12. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
* 13. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
* 14. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
* 15. Those who plan to donate ovum or sperms during the study period;
* 16. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
* 17. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of neutralizing antibodies against SARS-CoV-2 dominant epidemic variant on D14. | day 14 after the study vaccination
Seroresponse Rate (SRR) of neutralizing antibodies against SARS-CoV-2 dominant epidemic variant on D14. | day 14 after the study vaccination

SECONDARY OUTCOMES:
GMT of neutralizing antibodies against other SARS-CoV-2 variants on D14. | Day 14 after the study vaccination
SRR of neutralizing antibodies against other SARS-CoV-2 variants on D14. | Day 14 after the study vaccination
GMT and SRR of neutralizing antibodies against SARS-CoV-2 variants on D180. | day 14 after the study vaccination
Incidence and severity of solicited Adverse Events (AEs) of SCTV01E from D0 to D7. | Day 0 to Day 7 after the study vaccination
Incidence and severity of all unsolicited AEs of SCTV01E from D0 to D28. | Day 0 to Day 28 after the study vaccination
Incidence and severity of Serious Adverse Events (SAEs) and Adverse Event of Special Interests (AESIs) of SCTV01E within 365 days. | Day 0 to Day 180 after the study vaccination